CLINICAL TRIAL: NCT02349230
Title: The Effect of Astym Treatment on Acute Changes in Muscle Performance
Brief Title: The Effect of Astym Treatment on Muscle Performance
Acronym: Astym
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Responsible Party: Principal Investigator, Benjamin Kivlan, Instructor, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10Astym
Record Dates: First submitted 2015-01-19; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Musculoskeletal Pathology to the Lower Extremity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Astym treatment (Experimental): Astym treatment is a manual therapy intervention applied by certified therapists with specialized instruments
  Interventions: Other: Astym treatment
- Sham Astym (Sham Comparator): A sham Astym treatment applied with non-therapeutic pressure and
  Interventions: Other: Astym treatment
- Control (No Intervention): 12 minutes of rest

INTERVENTIONS:
Other: Astym treatment — Astym is a manual therapy technique applied by a certified therapist with advanced training in the technique. The technique is applied to a limb or body segment with specialized instruments in a specific sequential protocol that incorporates the muscle groups and joints of the entire kinetic chain.
  Arms: Astym treatment; Sham Astym

SUMMARY:
Subjects were randomized into 3 treatment groups (15 subjects per group): 1) Control - received no treatment 2) Placebo - received a sham Astym® treatment 3) Astym® Treatment - received Astym® treatment to the lower extremity. Subjects were blinded to whether they received the Astym® treatment or placebo treatment intervention. After a 5-minute warm-up on a lower body ergometer the subjects were familiarized to the operations of a computerized leg press machine that measured the maximum force output (Newtons) during a unilateral isometric squat test. A baseline measure of maximal force output (pre-test) was determined by the average of 3 trials with a 30 second rest period between the trials. The subjects then received the designated treatment intervention. Immediately following the treatment intervention (0 minutes following treatment intervention) the subjects were retested (post-test) using identical testing procedures by an investigator blinded to the treatment intervention received by the subject. Maximum force output measured in Newtons for the post-test was subtracted from the maximum force output (Newtons) pre-test and then converted to a percentage of change [(post-test - pretest)/pretest X 100). The percent change of maximal force output from pre-test to post-test measures was compared using a one-way analysis of variance with alpha set at 0.05. A Tukey's post-hoc analysis determined statistical differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Referral for physical therapy services to the student investigator for a musculoskeletal injury to the lower extremity.
2. Subjects must be aged between 18-65 years-old
3. Present with a 10% or greater deficit in maximum force output on computerized leg press machine when compared to the uninvolved side
4. Able to read and understand English language.
5. Read, comprehend, and sign informed consent procedures.

Exclusion Criteria:

1. Subjects who are pregnant
2. Subjects with a medical history of hemophilia or other clotting disorders of the blood
3. Subjects currently taking blood thinners (e.g. lovenox, Coumadin)
4. Subjects with neuropathy of the lower extremity
5. Subjects with a history of metastatic disease
6. Subjects with uncontrolled hypertension
7. Subjects that are unable to perform the strength test due to the nature of injury
8. Subjects with a recent history (within the past 4 weeks) of lower extremity surgery.
9. Subjects with compromised skin integrity. (e.g. open wounds, diabetic ulcers, lacerations, abrasions)
10. Subjects with any sign of infection including skin infections to the lower limbs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent Change in Maximal Force Output | Immediately following treatment intervention

REFERENCES:
- [Derived] Kivlan BR, Carcia CR, Clemente FR, Phelps AL, Martin RL. The effect of Astym(R) Therapy on muscle strength: a blinded, randomized, clinically controlled trial. BMC Musculoskelet Disord. 2015 Oct 29;16:325. doi: 10.1186/s12891-015-0778-9. PMID 26510526